CLINICAL TRIAL: NCT00964119
Title: An Interdisciplinary Study of Musculoskeletal Effects of Isotretinoin During Acne Treatment in Pediatric Population
Brief Title: Musculoskeletal Effects of Isotretinoin During Acne Treatment in Pediatric Population
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator has left Sponsoring Instiution
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2008-0106
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This is a prospective study, that will follow participants over their course of treatment on Isotretinoin. All patients who are prescribed Isotretinoin for their acne treatment are registered in iPLEDGE. The iPLEDGE program involves a set of steps that the patient, physician and pharmacist must follow for the patient to take Isotretinoin. Patients will be asked if they are willing to participate in this research study to determine musculoskeletal changes in adolescents and young adults on systemic therapy using the highly sensitive magnetic resonance (MR) imaging modality. In addition to the MRI, participants will be asked if they are willing to give an extra sample of blood when their routine blood work is being done for iPLEDGE. This blood sample will be used to determine if there are any effects of isotretinoin on bone turnover markers.

ELIGIBILITY:
Inclusion Criteria:

1. Registered in I-Pledge and has not started the Isotretinoin medication
2. Females and males ages 12-21 years old
3. Able to undergo 3 MRI scan

Exclusion Criteria:

1. Participants taking additional vitamin A, D or Calcium supplements
2. Previous musculoskeletal injuries (from incidental trauma, sports related injury or motorvehicle accidents, etc)
3. Clinical diagnosis of psoriasis, rheumatoid arthritis and/or Reiter's disease
4. relocation within the next 6 months
5. participation on a research study involving drug medication within the past 30 days

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All subjects will be recruited from the UW-Madison, Department of Dermatology located at 1 South Park Street, Madison, Wisconsin. Study flyers and brochures will be posted in the waiting areas and clinic rooms at the UW Dermatology clinics. UW Dermatologist will identify patients that meet study criteria and ask if they are interested in research participation, then they will be referred to study personnel for more information.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Teng, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Cohort Obervational
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Adolescents and young adults treated with systemic isotretinoin for recalcitrant inflammatory or nodular cystic acne.
Arm/Group | Single Cohort Observational
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Toxicities Related to the Use of Isotretinoin
Description: Bone Marker measurements to assess skeletal toxicities: Change in Bone specific Alkaline Phosphatase: (BSAP) over 5 months of therapy
Time Frame: Baseline to 5 months post therapy
Population: Pilot observational study; Principal Investigator left sponsoring institution, data analysis not completed. Data analysis based on interim data (12 subjects). No manuscript published. No final analysis expected. Study has been closed with the local IRB and files archived.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Single Cohort Observational
Number analyzed (Participants) | 12
U/L
  Baseline BSAP | 62.73 (35.86)
  post 5 month isotretinoin therapy | 51.80 (24.26)
Statistical Analysis 1: Comparison: Single Cohort Observational; PI and lead author left the institution before publishing data. Study has been closed and data files archived; Test type: Superiority or Other; p < .05, t-test, 2 sided — P-value < .05 is the computed p-value for this measurement

ADVERSE EVENTS:
Arm/Group | Single Cohort Observational
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Cohort Observational (N=15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) — (full body questionnaire)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes